CLINICAL TRIAL: NCT01797900
Title: Phase 2 Study of Inductive Plus Concurrent Chemoradiation Versus Concurrent Plus Adjuvant Chemoradiation for High-risk Locally Advanced Nasopharyngeal Carcinoma in the Era of IMRT
Brief Title: The Role of Induction Chemotherapy for High-risk Locally Advanced Nasopharyngeal Carcinoma in the Era of IMRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Li Gao, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-HN-002
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: adjuvants; inductive; concurrent; chemoradiotherapy; high-risk; locally advanced; NPC
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Cisplatin; Paclitaxel; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inductive + concurrent chemotherapy (Experimental): Inductive chemotherapy :paclitaxel 175mg/m2 d1+ cisplatin 80mg/m2d1, every 21 days for two cycles concurrent chemotherapy:cisplatin 80mg/m2 on week 1, 4, 7 radiotherapy: IMRT
  Interventions: Drug: Cisplatin; Drug: Paclitaxel; Radiation: IMRT
- concurrent + adjuvant chemotherapy (Active Comparator): concurrent chemotherapy: cisplatin 80 mg/m2, on week 1, 4, 7 adjuvant chemotherapy: paclitaxel 175mg/m2 + cisplatin 75mg/m2, every 21 days for 4 cycles radiotherapy: IMRT
  Interventions: Drug: Cisplatin; Drug: Paclitaxel; Radiation: IMRT

INTERVENTIONS:
Drug: Cisplatin — induction: Cisplatin: 80mg/m2, d1 and d22 concurrent: Cisplatin: 100mg/m2, d1, 22, 43 adjuvant: cisplatin: 75mg/m2, d1, d22, d43,d64
Drug: Paclitaxel — induction: paclitaxel 175mg/m2 d1,d22 adjuvant: paclitaxel 175mg/m2 d1,d22, d43,d64
Radiation: IMRT — 69.96Gy-73.43Gy to gross tumor volume, 60Gy to high-risk clinincal target volume, 50Gy to lower risk clincial target volume
  Other Names: intensity-modulated radiotherapy

SUMMARY:
The purpose of this study is to determine whether Intensity-modulated radiation therapy (IMRT) combined inductive and concurrent chemotherapy with more intensive regimen (cisplatin and paclitaxel) is feasible and effective than current standard treatment for high-risk locally advanced NPC patients.

DETAILED DESCRIPTION:
Meta-analysis showed chemotherapy when combined with conventional radiotherapy in locally advanced naso-pharyngeal carcinoma can improve 5-year overall survival with 6%, and beyond all concurrent chemotherapy with cisplatin benefits most. However, from Lin's (Lin JC, 2004) study, locally advanced NPC with high risk factors can not benefit from conventional concurrent chemoradiation. Failure pattern analysis revealed that local and distant failure accounted for 50% respectively. Large-scale data has demonstrated that with IMRT, local control can achieve 90%. Previous studies showed inductive chemotherapy can decrease distant metastasis. We need more effective and stronger chemotherapy, and we still need to testify concurrent chemotherapy combined with inductive chemotherapy.

A prospective trial would thus provide valuable information to help physicians and patients more precisely identify the feasibility and effectiveness of inductive + concurrent chemotherapy combined with IMRT for high-risk locally advanced NPC.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proved NPC
* N3 or T4N2 or multiple lymphnodes involved with at least one mass 4 cm or more in maximal diameter according to 7th UICC Staging
* provide written informed consent
* Kps>70
* no dostant metastasis
* Life expectancy≥6 months
* Adequate renal function, defined as follows: Serum creatinine < 2 x institutional upper limitof normal(ULN) within 2 weeks prior to registration or; creatinine clearance rate (CCr) ≥ 50 ml/min within 2 weeks prior to registration determined by 24- hour collection or estimated by Cockcroft-Gault formula: CCr male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dl) x (72)] CCr female = 0.85 x (CCrmale)
* The following assessments are required within 2 weeks prior to the start of registration: Na, K, Cl, glucose, Ca, Mg, and albumin.

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years; noninvasive cancers (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible) are permitted even if diagnosed and treated < 3 years ago
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Severe, active co-morbidity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Distant failure free survival | three years

SECONDARY OUTCOMES:
overall survival | three years
acute treatment toxicity | up to 16 weeks
late treatment toxicity | three years
Local recurrence rate | three years

CONTACTS AND LOCATIONS:
Overall Officials: Li Gao, MD, Study Director — Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China